CLINICAL TRIAL: NCT07339241
Title: Abdominal Circumference as a Novel Predictor of Operative Time in Retroperitoneal Adrenalectomy for Pheochromocytoma: A Retrospective Observational Study
Brief Title: Abdominal Circumference as a Predictor of Operative Time in Retroperitoneal Adrenalectomy for Pheochromocytoma
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Byung-Chang Kim, MD, PhD, Asan Medical Center
Other Study IDs: AC-PHEO-RPA
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pheochromocytoma Malignant
Keywords: Pheochromocytoma; retroperitoneal adrenalectomy; operative time; abdominal circumference
MeSH Terms: conditions — Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pheochromocytoma Patients: Patients diagnosed with pheochromocytoma who underwent retroperitoneal adrenalectomy at a single tertiary referral center. All procedures were performed as part of routine clinical care, and no experimental intervention was assigned for the purpose of this observational study.
  Interventions: Procedure: Retroperitoneal Adrenalectomy

INTERVENTIONS:
Procedure: Retroperitoneal Adrenalectomy — Retroperitoneal adrenalectomy performed as part of routine clinical care for patients with pheochromocytoma. No experimental intervention was assigned, and the surgical procedure was not altered for the purpose of this observational retrospective study.

SUMMARY:
This retrospective observational study examines whether abdominal circumference is associated with operative time in patients undergoing retroperitoneal adrenalectomy for pheochromocytoma. Data were collected from medical records of patients treated at a single tertiary referral center. The primary outcome is operative time, measured in minutes. The purpose of this study is to evaluate whether abdominal circumference can serve as a practical predictor of operative difficulty in retroperitoneal adrenalectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with pheochromocytoma
* Patients who underwent retroperitoneal adrenalectomy
* Availability of complete operative records

Exclusion Criteria:

* Patients younger than 18 years
* Patients who underwent transperitoneal adrenalectomy
* Incomplete clinical or operative data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with pheochromocytoma who underwent retroperitoneal adrenalectomy at a single tertiary referral center. Data were collected retrospectively from electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Operative Time | During surgery
  Operative time measured in minutes from skin incision to skin closure, obtained from operative records.

CONTACTS AND LOCATIONS:
Overall Officials: BYUNG-CHANG KIM, MD, PhD, Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No